CLINICAL TRIAL: NCT00846183
Title: Effect of Local Injury to Endometrium on the Day of Oocyte Retrieval in First IVF Cycle on Implantation Rate.
Brief Title: Effect of Local Injury on Implantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yazd Research & Clinical Center for Infertility (Other)
Responsible Party: Principal Investigator, homa oskouian, fellowship, Yazd Research & Clinical Center for Infertility
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: local injury111
Record Dates: First submitted 2009-02-17; First posted 2009-02-18 (Estimated); Last update posted 2013-12-23 (Estimated); Status verified 2013-12

CONDITIONS: Implantation Rate
Keywords: local injury; implantation rate; endometrial receptivity; IVF

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- local ingury (Active Comparator): In one group, on the day of oocyte retrieval, local injury to endometrium with a Novak curet to anterior and posterior wall of endometrium are performed.
  Interventions: Procedure: local injury
- control (No Intervention): in 60 patients routine IVF are performed

INTERVENTIONS:
Procedure: local injury — In one group, on the day of oocyte retrieval, local injury to endometrium with a Novak curet to anterior and posterior wall of endometrium are performed
  Other Names: it does not have other name
  Arms: local ingury

SUMMARY:
Local injury on two sights of endometrium are performed in 60 patients in their first IVF cycle and implantation rate are compared with fresh cycles without local injury.

DETAILED DESCRIPTION:
Low implantation rate is still a major concern in ART cycles. It has been reported that local injury to endometrium may improve endometrial receptivity and implantation rate. A total of 120 patients in first IVF cycles, who are stimulated with long protocol, are randomly divided into two groups. In one group, on the day of oocyte retrieval, local injury to endometrium with a Novak curet to anterior and posterior wall of endometrium are performed and in the other group no interventions are done. After fresh embryo transfers, implantation and clinical pregnancy rates are compared between two groups.

ELIGIBILITY:
Inclusion Criteria:

* Age < 35
* First IVF cycle
* Long protocol should be used for stimulation

Exclusion Criteria:

* Day 3 FSH > 10

Max Age: 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 156 (Actual)
Dates: Start 2008-06; Primary Completion 2008-11 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
implantation rate | 4 weeks

SECONDARY OUTCOMES:
clinical pregnancy rate | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: homa oskouian, M.D., Principal Investigator — Research and clinical center for infertility; Mohamad ali karimzade, MD, Principal Investigator — Research and clinical center for infertility
Locations (1):
- Research and clinical center for infertility, Yazd, Yazd Province, Iran

REFERENCES:
- [Derived] Lensen SF, Armstrong S, Gibreel A, Nastri CO, Raine-Fenning N, Martins WP. Endometrial injury in women undergoing in vitro fertilisation (IVF). Cochrane Database Syst Rev. 2021 Jun 10;6(6):CD009517. doi: 10.1002/14651858.CD009517.pub4. PMID 34110001